CLINICAL TRIAL: NCT00697255
Title: A Phase II, Randomized, Controlled, Open-label, Feasibility Trial to Evaluate if a Single or Repeated Dose of Org 36286 (Corifollitropin Alfa) Followed by a Low Daily Dose of Either hCG or Recombinant FSH Can Induce Monofollicular Growth in Women With WHO Group II Anovulatory Infertility
Brief Title: A Phase 2 Trial to Evaluate if Corifollitropin Alfa (Org 36286), Followed by a Low Daily Dose of hCG or Recombinant FSH Can Induce Monofollicular Growth in Women With WHO Group II Anovulatory Infertility (P05693)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05693; 2006-000705-30 (EudraCT Number); 107010 (Other: Organon); MK-8962-002 (Other: Merck)
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2022-02

CONDITIONS: Ovulation Induction
Keywords: Pharmacological effects of drugs; Hormones; Hormone Substitutes and Hormone Antagonists; Pharmacological Actions; Monofollicular growth; Randomized; Open-label; Active-controlled
MeSH Terms: interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; Glycoprotein Hormones, alpha Subunit; follitropin beta; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- corifollitropin alfa + recFSH (Experimental): Eligible participants will receive a subcutaneous (SC) injection of corifollitropin alfa (Stage 1a: 15mcg, Stage Ib/II: 30 mcg) the first, second, or third day after onset of a progestagen-induced withdrawal bleeding. If the follicle growth is insufficient, the participant will receive a second or third dose of corifollitropin alfa (Stage 1a: 15 mcg, Stage Ib/II: 20 mcg). As soon as the largest follicle reaches a size of ≥12 mm, the participant will start daily SC injections with FSH (Stage 1A: 50 IU, Stage II: 75 IU) the same day. A bolus injection of hCG (5000 IU) will be administered if at least one follicle is ≥18 mm and in total no more than two follicles ≥15 mm are observed.
  Interventions: Drug: corifollitropin alfa; Biological: recombinant Follicle Stimulating Hormone (recFSH); Biological: hCG Bolus injection
- corifollitropin alfa + hCG (Experimental): Eligible participants will receive a SC injection of corifollitropin alfa (Stage Ia:15 mcg, Stage Ib/II: 30 mcg) the first, second or third day after onset of a progestagen-induced withdrawal bleeding. If the follicle growth is insufficient the participant will receive a second or third dose of corifollitropin alfa (Stage IA: 15 mcg, stage Ib/II: 20 mcg). As soon as the largest follicle reaches a size of ≥12 mm the participant will start daily SC injections with hCG (Stage Ib/II: 200 IU) the same day. A bolus injection of hCG (5000 IU) will be administered if at least one follicle is ≥18 mm and in total no more than two follicles ≥15 mm are observed.
  Interventions: Drug: corifollitropin alfa; Biological: human Chorion Gonadotropin (hCG); Biological: hCG Bolus injection

INTERVENTIONS:
Drug: corifollitropin alfa — SC corifollitropin alfa on the 1st, 2nd or 3rd day after onset of a progestagen-induced withdrawal bleeding (Stage 1a: 15mcg, Stage Ib/II: 30 mcg).
  Other Names: Org 36286; SCH 900962; MK-8962
Biological: recombinant Follicle Stimulating Hormone (recFSH) — Daily injections of SC recFSH (50 IU/75 IU) administered as soon as the largest follicle reaches a size ≥12 mm 4 days after a corifollitropin alfa injection on stimulation day 5, 9 or 13.
  Other Names: Puregon®
  Arms: corifollitropin alfa + recFSH
Biological: human Chorion Gonadotropin (hCG) — Daily injections of SC hCG (200 IU) administered as soon as the largest follicle reaches a size ≥12 mm 4 days after a corifollitropin alfa injection on stimulation day 5, 9 or 13.
  Other Names: Pregnyl®
  Arms: corifollitropin alfa + hCG
Biological: hCG Bolus injection — Bolus injection of SC hCG was administered to induce final oocyte maturation if at least one follicle is ≥18 mm and no more than two follicles ≥15 mm are observed.
  Other Names: Pregnyl®

SUMMARY:
The primary objective of this trial is to evaluate whether a corifollitropin alfa (Org 36286) regimen applying a single or repeated dose of corifollitropin alfa followed by a low daily dose of Human Chorion Gonadotropin (hCG) or recombinant Follicular Stimulating Hormone (recFSH) can induce monofollicular growth (one follicle ≥18 mm and no other follicle ≥15 mm at day of bolus injection of hCG) in women with WHO group II anovulatory infertility.

DETAILED DESCRIPTION:
This trial will include two separate stages (Ia+Ib and II).

Stage Ia will be open-label and uncontrolled in a small cohort of women (n=5) to explore whether the intended dosing regimen of corifollitropin alfa followed by daily low dose recFSH provide an appropriate response in eligible participants meeting all inclusion and none of the exclusion criteria.

Stage Ib will be open-label and uncontrolled in a small cohort of women (n=5) to explore whether the intended dosing regimen of corifollitropin alfa followed by daily low dose hCG provide an appropriate response in eligible participants meeting all inclusion and none of the exclusion criteria.

Stage II is open-label and randomized (n=40) to evaluate whether the intended dosing regimen of corifollitropin alfa followed by low dose FSH (n=20) or hCG (n=20) provide an appropriate response in eligible participants meeting all inclusion and none of the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Oligomenorrhea (average cycle length ≥35 days and <6 months)
* Amenorrhea (average cycle length ≥6 months)
* Body Mass Index ≥18 and ≤30 kg/m^2
* Normal serum FSH levels and normal estradiol levels at screening
* Progestagen induced withdrawal bleeding
* Age ≥18 years and ≤39 years at the time of signing informed consent
* Willing and able to sign informed consent

Exclusion Criteria:

* History of or current ovarian cysts or enlarged ovaries not related to polycystic ovarian syndrome (PCOS)
* History of or current tumors of the ovary, breast, uterus, pituitary or

hypothalamus

* Less than 2 ovaries
* Undiagnosed vaginal bleeding
* Any ovarian and/or abdominal abnormality interfering with ultrasound

examination

* Malformations of the sexual organs incompatible with pregnancy
* Pregnancy or lactation
* Abnormal serum endocrinology levels based on screening sample
* Any clinically relevant abnormal laboratory value based on screening sample
* Alcohol or drug abuse within the 12 months preceding signing of informed consent
* Hypersensitivity to any of the substances in corifollitropin alfa
* Hypersensitivity to hCG/ Puregon® or any of its components
* Previous use of corifollitropin alfa
* Use of any investigational drug during 90 days before screening

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2007-05-15 (Actual); Primary Completion 2008-04-03 (Actual); Study Completion 2008-05-15 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants were enrolled in Stage 1a to receive corifollitropin alfa + recombinant Follicular Stimulating Hormone (recFSH), and 3 participants were enrolled in Stage 1b to receive corifollitropin alfa + Human Chorion Gonadotropin (hCG).
Groups:
- Corifollitropin Alfa + recFSH: Eligible participants in Stage 1a received a subcutaneous (SC) injection of corifollitropin alfa (15 mcg) the first, second, or third day after onset of a progestagen-induced withdrawal bleeding. If the follicle growth was insufficient, the participant received a second or third dose of corifollitropin alfa (15 mcg). As soon as the largest follicle reached a size of ≥12 mm, the participant started daily SC injections with recFSH (50 IU) the same day. A bolus injection of hCG (5000 IU) was administered if at least one follicle was ≥18 mm and in total no more than two follicles ≥15 mm were observed.
- Corifollitropin Alfa + hCG: Eligible participants in Stage 1b received a SC injection of corifollitropin alfa (30 mcg) the first, second or third day after onset of a progestagen-induced withdrawal bleeding. If the follicle growth was insufficient the participant received a second or third dose of corifollitropin alfa (20 mcg). As soon as the largest follicle reached a size of ≥12 mm the participant started daily SC injections with hCG (200 IU) the same day. A bolus injection of hCG (5000 IU) was administered if at least one follicle was ≥18 mm and in total no more than two follicles ≥15 mm were observed.
Period: Stage 1a
Arm/Group | Corifollitropin Alfa + recFSH | Corifollitropin Alfa + hCG
Started | 5 | 0
Completed | 2 (Participants who completed 1a received hCG bolus injection and did not proceed further in the trial) | 0
Not Completed | 3 | 0
Not completed — Insufficient ovarian response | 1 | 0
Not completed — Multifollicular growth | 1 | 0
Not completed — Not growing of dominant follicle | 1 | 0
Period: Stage 1b
Arm/Group | Corifollitropin Alfa + recFSH | Corifollitropin Alfa + hCG
Started | 0 | 3 (After enrollment in Stage 1a completed, a new cohort of participants enrolled in Stage 1b.)
Completed | 0 | 1 (Participants who completed 1b received hCG bolus injection and did not proceed further in the trial)
Not Completed | 0 | 2
Not completed — Not growing of dominant follicle | 0 | 1
Not completed — Insufficient ovarian response | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Corifollitropin Alfa + recFSH | Corifollitropin Alfa + hCG | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (5.9) | 28.7 (2.5) | 30.0 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Monofollicular Response (Monofollicular Rate)
Description: The monofollicular rate was defined as the number of participants with monofollicular response (one follicle ≥18 mm and no other follicle ≥15 mm on the day of the bolus injection of hCG) divided by the number of the treated participants.
Time Frame: At day of bolus injection of hCG (up to 20 days)
Population: Intent-to-Treat group (ITT) consisted of all treated participants (5 participants in Stage Ia and 3 participants in Stage Ib).
Measure: Number; unit: percentage of participants
Arm/Group | Corifollitropin Alfa + recFSH | Corifollitropin Alfa + hCG
Number analyzed (Participants) | 5 | 3
percentage of participants | 0 | 0

2. Secondary Outcome: Percentage of Participants With Ovulation (Ovulation Rate)
Description: Ovulation rate was defined as the number of participants with confirmed ovulation (≥15 nmol/l serum progesterone eight days after the bolus injection of hCG) divided by the number of treated participants. Ovulation was also considered confirmed for participants who became pregnant, had an ectopic pregnancy or had a miscarriage.
Time Frame: 8 days after bolus injection of hCG (up to 28 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Corifollitropin Alfa + recFSH | Corifollitropin Alfa + hCG
Number analyzed (Participants) | 5 | 3
percentage of participants | 40.0 | 33.3

3. Secondary Outcome: Percentage of Participants With Monofollicular Ovulation (Monofollicular Ovulation Rate)
Description: Monofollicular ovulation rate was defined as the number of participants with monofollicular response (one follicle ≥18 mm and no other follicle ≥15 mm on the day of the bolus injection of hCG) and confirmed ovulation (≥15 nmol/l serum progesterone eight days after the bolus injection of hCG) divided by the number of treated participants. Ovulation was also considered confirmed for participants who became pregnant, had an ectopic pregnancy or had a miscarriage.
Time Frame: 8 days after bolus injection of hCG (up to 28 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Corifollitropin Alfa + recFSH | Corifollitropin Alfa + hCG
Number analyzed (Participants) | 5 | 3
percentage of participants | 0 | 0

4. Secondary Outcome: Percentage of Participants Who Cancelled Treatment (Cancellation Rate)
Description: Treatment was considered cancelled if no bolus injection of hCG was administrated. Reasons of treatment failure included Adverse Event (AE)/ Serious Adverse Event (SAE), insufficient ovarian response on stimulation day 13 (no follicle ≥12 mm), insufficient ovarian response after 7 days of hCG/recFSH treatment (no follicle ≥18 mm), and multifollicular growth (≥3 follicles ≥15 mm).
Time Frame: Up to 3 weeks after bolus injection of hCG (up to 41 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Corifollitropin Alfa + recFSH | Corifollitropin Alfa + hCG
Number analyzed (Participants) | 5 | 3
percentage of participants
  Insufficient ovarian response | 20.0 | 33.3
  Multifollicular growth | 20.0 | 0
  Not growing of dominant follicle | 20.0 | 33.3

5. Secondary Outcome: Number of Participants With Pregnancy
Description: A pregnancy test (serum or urinary hCG) was performed two to three weeks after bolus injection of hCG. In case of a positive pregnancy test vaginal and/or abdominal ultrasound scan was performed to confirm the pregnancy at 5 to 6 weeks after bolus injection of hCG and ≥10 weeks after bolus injection of hCG to confirm ongoing pregnancy.
Time Frame: At least 10 weeks after bolus injection of hCG (up to 13 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa + recFSH | Corifollitropin Alfa + hCG
Number analyzed (Participants) | 5 | 3
participants | 0 | 1

6. Secondary Outcome: Number of Participants With AEs of Ovarian Hyperstimulation Syndrome (OHSS)
Description: OHSS was classified on study based on a slightly modified WHO Scientific Group (1973) classification: Grade I (mild) = characterized by excessive steroid secretion and ovarian enlargement (5-7 cm). Abdominal discomfort, including abdominal pain, is present. Grade II (moderate) = characterized by distinct ovarian cysts (ovary size 8-10 cm), accompanied by abdominal pain and tension, nausea, vomiting, diarrhea. Grade III (severe) = characterized by enlarged cystic ovaries (ovary size >10 cm), accompanied by ascites and occasionally hydrothorax. Abdominal tension and pain may be severe. Pronounced hydrothorax together with an abdominal cavity filled with cysts and fluid elevating the diaphragm may cause severe breathing difficulties. Large quantities of fluid inside the cysts and in the peritoneal and pleural cavities cause haemoconcentration and increased blood viscosity. In rare cases, the syndrome may further be complicated by the occurrence of thromboembolic phenomena.
Time Frame: During In-Treatment Period (up to 14 weeks after first corifollitropin injection)
Population: The All-Participants-Treated (APT) group consisted of all participants who received corifollitropin alfa. Participants were grouped according to the stage of the trial and the active treatment group (recFSH Stage Ia, hCG Stage Ib) they actually received.
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa + recFSH | Corifollitropin Alfa + hCG
Number analyzed (Participants) | 5 | 3
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: During In-Treatment Period (up to 14 weeks after first corifollitropin injection)
Arm/Group | Corifollitropin Alfa + recFSH | Corifollitropin Alfa + hCG
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 2/5 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corifollitropin Alfa + recFSH (N=5) | Corifollitropin Alfa + hCG (N=3)
Listless (Psychiatric disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications must be based on data validated and released by the Sponsor. Any such scientific paper, presentation, or other communication concerning the clinical trial described in the protocol will first be submitted to the Sponsor, at least 6 weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.